CLINICAL TRIAL: NCT02746575
Title: Novel Strategy For Perioperative Beta-Blocker Therapy - Pilot Study
Brief Title: Pilot - Peri-operative Beta Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201507010
Record Dates: First submitted 2016-04-14; First posted 2016-04-21 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Adrenergic Beta-Receptor Blockader; Troponin Levels; Cardiomyopathy, Post-surgical
MeSH Terms: conditions — Cardiomyopathies | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): Postsurgical: 5mg metoprolol, IV, prior to extubation, every 5 minutes to achieve target heart rate of 65/min, up to 15mg; then 25mg metoprolol, oral, every 8 hours for 72 hours.
  Interventions: Drug: metoprolol

INTERVENTIONS:
Drug: metoprolol
  Other Names: Lopressor

SUMMARY:
Perioperative cardiac adverse events [heart injuries caused by general anesthesia and surgical procedures] are a significant public health issue, with more than 60,000 deaths per annum in patients having surgery for non-heart related issues. There are virtually no evidence-based medical strategies for effective prevention of these events. Preoperative drug treatment with beta blockade drugs used for high blood pressure, perioperative therapy with lipid lowering drugs such as statins, alpha-receptor agonists such as clonidine used for high blood pressure, and aspirin have all been investigated as potential mitigating treatments, but without positive clinical outcomes and, in some cases, creating more hemodynamic instabilities that result in heart injury. In light of this, investigators propose to evaluate the safety and efficacy of using increasing doses of beta blockade drugs immediately after surgery and to assess the value of high-sensitivity cardiac troponin level testing of the blood in predicting those patients who would benefit most from perioperative beta blocker therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years
* American Society of Anesthesiologists (ASA) risk status III-IV
* Revised Cardiac Risk Index ≥2
* β-blocker naïve (not having received β-blocker within 30 days prior to surgery)
* Previously diagnosed coronary artery disease (CAD) or at high risk for CAD:
* History of peripheral vascular disease, or
* Diabetes and currently on oral anti-diabetic drug or insulin therapy, or
* Chronic renal failure (eGFR <30 m/min)
* Major non-cardiac surgery under general anesthesia

Exclusion Criteria:

* History of stroke
* Heart rate <55bpm
* Heart failure
* Second or third degree AV block without pacemaker
* Active asthma or COPD
* Anemia [Hb<9g/dL]
* Allergy to beta-blockade drugs
* Hemodynamic instability
* Uncontrolled hemorrhage
* Unwilling or unable to give consent for participation

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes-Jewish Hospital/Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Postsurgical: 5mg metoprolol, IV, prior to extubation, every 5 minutes to achieve target heart rate of 65/min, up to 15mg; then 25mg metoprolol, oral, every 8 hours for 72 hours.
  metoprolol
Period: Overall Study
Arm/Group | Treatment
Started | 70
Completed | 20
Not Completed | 50
Not completed — Surgery cancelled or time chaned | 13
Not completed — Received epidural | 10
Not completed — Withdrawal by Subject | 3
Not completed — Bradycardia/hypotension | 9
Not completed — Study paused | 8
Not completed — put on beta-blocker | 3
Not completed — type of surgery | 1
Not completed — typ of surgery | 1
Not completed — PI unavailable | 1
Not completed — Unknown history of CVA | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Difference in hscTnI Values
Description: Difference in hscTnI concentrations between preoperative clinic visit and day of surgery
Time Frame: Before surgery and Immediately after surgery (on the day of surgery)
Population: Only patients with complete hscTnI data were inlcuded
Measure: Median (Inter-Quartile Range); unit: ng/L
Arm/Group | Treatment
Number analyzed (Participants) | 18
ng/L
  Preoperative visit | 3.4 [2.0 to 4.8]
  Day of surgery | 2.8 [2.3 to 4.4]

ADVERSE EVENTS:
Time Frame: Day of surgery until postoperative day 3 or hospital discharge
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT02746575/Prot_SAP_000.pdf